CLINICAL TRIAL: NCT01180660
Title: The Effect of Systemic Intraoperative Lidocaine on Postoperative Pain and Quality of Recovery on Morbid Obese Patients Undergoing Laparoscopic Gastric Bypass Surgery
Brief Title: IV Lidocaine on Postoperative Pain and QOR on Morbid Obese Patients Undergoing Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00032300
Record Dates: First submitted 2010-07-19; First posted 2010-08-12 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Pain; Obesity
Keywords: Gastric Surgery; Pain; Recovery; Laparoscopic Surgery
MeSH Terms: conditions — Pain; Obesity | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine infusion
  Interventions: Drug: Lidocaine Infusion
- Placebo (Placebo Comparator): Placebo Normal Saline Infusion
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine Infusion — 1.5 mg/kg bolus followed by an infusion of 2 mg/kg/hr throughout the intra operative period
  Arms: Lidocaine
Drug: Normal Saline — Saline bolus equal to that of lidocaine in addition to continuous infusion of normal saline during the intra operative period
  Other Names: Placebo infusion
  Arms: Placebo

SUMMARY:
Can Intraoperative systemic lidocaine decrease postoperative opioid consumption and improve quality of recovery after laparoscopic gastric bypass surgery? The hypotheses:does the use of intraoperative systemic lidocaine decrease postoperative opioid consumption and improve quality of recovery after laparoscopic gastric bypass surgery.

This study has the potential to confirm an opioid sparing strategy for morbid obese patients undergoing laparoscopic gastric bypass surgery. The high incidence of obstructive sleep apnea and the increased risk of postoperative hypoxemia make the development of opioid sparing techniques in this patient population warranted.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II,III;
* BMI > 35 kg/m2,
* Age between 18-70,
* Fluent in English,
* Patients undergoing laparoscopic gastric bypass,
* EKG within 3 months.

Exclusion Criteria:

* History of allergy to local anesthetics,
* History of chronic opioid use,
* Pregnant patients,
* History of EKG abnormalities.

Dropout: Conversion to open, patient or surgeon request.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, M.D, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Mun EC, Blackburn GL, Matthews JB. Current status of medical and surgical therapy for obesity. Gastroenterology. 2001 Feb;120(3):669-81. doi: 10.1053/gast.2001.22430. PMID 11179243
- [Background] Peiser J, Lavie P, Ovnat A, Charuzi I. Sleep apnea syndrome in the morbidly obese as an indication for weight reduction surgery. Ann Surg. 1984 Jan;199(1):112-5. doi: 10.1097/00000658-198401000-00020. PMID 6691724
- [Background] Kyzer S, Charuzi I. Obstructive sleep apnea in the obese. World J Surg. 1998 Sep;22(9):998-1001. doi: 10.1007/s002689900506. PMID 9717428
- [Background] Rosenberg-Adamsen S, Kehlet H, Dodds C, Rosenberg J. Postoperative sleep disturbances: mechanisms and clinical implications. Br J Anaesth. 1996 Apr;76(4):552-9. doi: 10.1093/bja/76.4.552. No abstract available. PMID 8652329
- [Background] Alexander CM, Gross JB. Sedative doses of midazolam depress hypoxic ventilatory responses in humans. Anesth Analg. 1988 Apr;67(4):377-82. PMID 3354874
- [Background] Wills VL, Hunt DR. Pain after laparoscopic cholecystectomy. Br J Surg. 2000 Mar;87(3):273-84. doi: 10.1046/j.1365-2168.2000.01374.x. PMID 10718794
- [Background] Goldstein A, Grimault P, Henique A, Keller M, Fortin A, Darai E. Preventing postoperative pain by local anesthetic instillation after laparoscopic gynecologic surgery: a placebo-controlled comparison of bupivacaine and ropivacaine. Anesth Analg. 2000 Aug;91(2):403-7. doi: 10.1097/00000539-200008000-00032. PMID 10910857
- [Background] Shaw IC, Stevens J, Krishnamurthy S. The influence of intraperitoneal bupivacaine on pain following major laparoscopic gynaecological procedures. Anaesthesia. 2001 Nov;56(11):1041-4. doi: 10.1046/j.1365-2044.2001.02215.x. PMID 11703235
- [Background] Moiniche S, Mikkelsen S, Wetterslev J, Dahl JB. A qualitative systematic review of incisional local anaesthesia for postoperative pain relief after abdominal operations. Br J Anaesth. 1998 Sep;81(3):377-83. doi: 10.1093/bja/81.3.377. PMID 9861124

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 subjects were randomized and 50 completed the study. Subjects were enrolled consecutively from August 2010 through October 2012.
Pre-assignment Details: 60 subjects were assessed for eligibility and 9 were excluded because they did not meet inclusion criteria n=3 or the subject refused n=6.
  51 subjects were randomized to the study
Period: Overall Study
Arm/Group | Lidocaine | Placebo
Started | 25 | 26
Completed | 24 | 26
Not Completed | 1 | 0
Not completed — Changed to open surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Placebo | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 51
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51
Body Mass Index [Median (Inter-Quartile Range); unit: Unit of measure (kg/m2)] | 47 [42 to 54] | 48 [44 to 53] | 47 [43 to 53]

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery 40 on the Day After Surgery
Description: Quality of Recovery 40 on the Day After Surgery. The survey is a quality of recovery tool and a score of 40 is low and 200 is high.
  The minimum score is 40 which is minimum recovery score and them maximum score is 200 which is considered better recovery.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on scale 40 (low) - 200 (high)
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 24 | 26
units on scale 40 (low) - 200 (high) | 165 [151 to 170] | 146 [130 to 169]
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; A sample size of 22 subjects per group was estimated to achieve 90% power to detect a 16 point difference in the aggregated Qor-40 score for the two study groups to be compared assuming an overall standard deviation of 16 points similar to what was observed in a previous investigation; Test type: Superiority or Other; p = .01, Regression, Linear; Median Difference (Net) = 19, 95% CI 2-sided [3 to 27]

2. Secondary Outcome: 24 Hour Total Opioid Consumption
Description: 24 hour total opioid consumption using IV morphine equivalents
Time Frame: 24 hours post surgery
Measure: Median (Inter-Quartile Range); unit: miligrams
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 24 | 26
miligrams | 26 [19 to 46] | 36 [24 to 65]

ADVERSE EVENTS:
Time Frame: 24 hours after surgery
Arm/Group | Lidocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 5/24 | 14/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=24) | Placebo (N=26)
Nausea (Gastrointestinal disorders) | 5 (5) | 14 (14) — Nausea

LIMITATIONS AND CAVEATS:
We did not evaluate if the opioid sparing properties of systemic lidocaine resulted in a lower incidence of adverse respiratory events (hypoxemia/hypoventilation). We were underpowered to detect significant differences in certain parts of the qor-40.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No